CLINICAL TRIAL: NCT02727400
Title: Impact on Mitochondrial Energy Production in Different Patient Populations in Women Undergoing IVF-ICSI (in Vitro Fertilization-intracytoplasmic Sperm Injection)
Brief Title: Mitochondrial Energy Production in ART (Assisted Reproductive Technology )
Acronym: Mitenergy
Status: Completed | Type: Observational
Sponsor: IVI Madrid (Other)
Responsible Party: Sponsor
Other Study IDs: 1512-MAD-064-JGPROTOCOLOf-151
Record Dates: First submitted 2016-01-23; First posted 2016-04-04 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Female Infertility Due to Advanced Maternal Age

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum, follicular fluid and granulosa cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- advanced maternal age: Infertile women due to advanced maternal age
- Young patients: women under 35 undergoing infertility treatments

SUMMARY:
Oocyte maturation requires a lot of energy, which is provided by the mitochondria via the synthesis of ATP. The majority of patients with advanced maternal age (AMA) have poor egg quality. One of the reasons depends on oxidative phosphorylation of Pyruvate to undergo maturation; on the contrary, the cells of the cumulus (CC) show great activity glycolytic so that these cells are able to provide ATP(adenosine triphosphate and energy substrates to the oocyte. The goal of this work is to analyze the mitochondrial function and energy production in oocyte donors compared with a group of women of advanced maternal age subject to a same ovarian stimulation Protocol

ELIGIBILITY:
Inclusion Criteria:

* Controls: Women between 18-35 years old who are oocyte donors and fulfill the requirements of the our program of oocyte donation according to the Spanish Law of Human Reproduction
* Cases: infertile women undergoing IVF due to advanced maternal age (>38 years)

Exclusion criteria:

For controls: Women with antral follicle count >20 or <6 follicle per ovary or with pathologies which, in the opinion of the investigator, may interfere with the treatment of ovarian stimulation

* Severe hypersensitivity to drugs of similar structure
* In the case of associated pathologies which can be considered as exclusion criteria on the part of the researcher are endocrine disruption and multi-follicular ovaries with risk of OHSS (Ovarian hyperstimulation syndrome)
* Be positive in serology for syphilis, toxoplasmosis, rubella, gonorrhea, hepatitis B, hepatitis C and HIV and lack of personal history and family of hereditary diseases.

Cases

* Irregular cycles
* Previous Ovarian surgery
* Previous chemotherapy or radiotherapy

Ages: 18 Years to 46 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Controls: Young women between 18-35 years old with good reproductive prognostic undergoing COS (controlled ovarian stimulation) for IVF-ICSI
  Cases: Infertile Women > 38 years old undergoing COS (controlled ovarian stimulation) for IVF-ICSI
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-04-16 (Actual); Study Completion 2018-04-16 (Actual)

PRIMARY OUTCOMES:
Adenosine Triphosphate (ATP) production (nmol) | 15 days
  ATP levels with the ATP assay kit (ab113849) Succinate dehydrogenase (SDH) activity assay kit (BioVision, USA) Mitochondrial Complex IV by colorimetric determination of oxidation-reduction processes of Cytochrome C

CONTACTS AND LOCATIONS:
Overall Officials: Juan A Garcia-Velasco, MD, PhD, Principal Investigator — IVI Madrid
Locations (1):
- IVI Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No